CLINICAL TRIAL: NCT00830947
Title: The OrthoAccel (OATI) Celerect Device Pivotal Study - Effect of Cyclic Loading (Vibration) on Orthodontic Tooth Movement
Brief Title: Effect of Cyclic Loading (Vibration) on Orthodontic Tooth Movement
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: OrthoAccel Technologies Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OA-02
Record Dates: First submitted 2009-01-26; First posted 2009-01-28 (Estimated); Results first posted 2013-12-23 (Estimated); Last update posted 2013-12-23 (Estimated); Status verified 2013-11

CONDITIONS: Malocclusion
Keywords: Orthodontic; Extraction; Device; Space Closure; Orthodontic malocclusion
MeSH Terms: conditions — Malocclusion

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- OrthoAccel Device (Experimental): Device provides a light vibration at 0.25 Newtons and 30 Hz frequency for 20 minutes daily.
  Interventions: Device: OrthoAccel Device
- Sham Device (inactive device) (Sham Comparator): Sham device will look identical to active devices but will not deliver vibration to the patient.
  Interventions: Device: Sham Device

INTERVENTIONS:
Device: OrthoAccel Device — The OA device provides a light vibration at 0.25 Newtons and 30 Hz frequency for 20 minutes daily.
  Arms: OrthoAccel Device
Device: Sham Device — Inactive sham device that is held in the mouth for 20 minutes.
  Arms: Sham Device (inactive device)

SUMMARY:
To gather data indicating whether or not the OrthoAccel device speeds tooth movement in people who use orthodontics (braces).

DETAILED DESCRIPTION:
This is a randomized, blinded study that will follow 32 patients for up to six months. Patients will have a minimum of 3 mm of extraction space that needs to be closed by moving the anterior teeth or canine distally. Patients will have standard orthodontic treatment and temporary anchorage devices for tooth movement and space closure. Half the patients will receive a functioning device and half the patients will receive a sham-device. Patients will use the device for 20 minutes daily; the device has a mouthpiece for the patient to lightly bite into plus a connected enclosure that stays outside the mouth. The enclosure provides a light vibration.

ELIGIBILITY:
Inclusion Criteria:

* Permanent dentition between the ages of 12 and 40
* Minimum of 3 mm of extraction space to be closed by distal movement of all 6 anterior teeth from canine to canine or by distal movement of the canines
* Good oral hygiene and compliance

Exclusion Criteria:

* Any compromised medical or dental condition
* Patient currently involved in any other study
* Lives significantly outside San Antonio, TX
* use of bisphosphonates
* pregnant females

Ages: 12 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 45 (Actual)
Dates: Start 2009-02; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Gakunga, DDS, Principal Investigator — University of Texas Health Science Center San Antonio
Locations (1):
- Ravi Anthony, San Antonio, Texas, United States

REFERENCES:
- [Derived] El-Angbawi A, McIntyre G, Fleming PS, Bearn D. Non-surgical adjunctive interventions for accelerating tooth movement in patients undergoing orthodontic treatment. Cochrane Database Syst Rev. 2023 Jun 20;6(6):CD010887. doi: 10.1002/14651858.CD010887.pub3. PMID 37339352

RESULTS

PARTICIPANT FLOW:
Groups:
- OrthoAccel Device: OrthoAccel Device : The OA device provides a light vibration at 0.2 Newtons and 30 Hz. frequency for 20 minutes daily.
- Sham (Inactive Device): Sham Device : Inactive sham device that is held in the mouth for 20 minutes.
Period: Overall Study
Arm/Group | OrthoAccel Device | Sham (Inactive Device)
Started | 23 | 22
Completed | 19 | 18
Not Completed | 4 | 4
Not completed — Lost to Follow-up | 4 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | OrthoAccel Device | Sham (Inactive Device) | Total
Number analyzed (Participants) | 23 | 22 | 45
Age Continuous [Mean (Standard Deviation); unit: years] | 21.8 (8.7) | 21.4 (7.8) | 21.6 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 11 | 28
  Male | 6 | 11 | 17

OUTCOME MEASURES:

1. Primary Outcome: The Rate of Orthodontic Movement of a Maxillary Canine Tooth Being Distalized to Close an Extraction Space.
Time Frame: Time to Space Closure, an average of 22 weeks
Measure: Mean (Standard Deviation); unit: mm/week
Arm/Group | OrthoAccel Device | Sham (Inactive Device)
Number analyzed (Participants) | 23 | 22
mm/week | 0.27 (0.04) | 0.18 (0.04)

ADVERSE EVENTS:
Arm/Group | OrthoAccel Device | Sham (Inactive Device)
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/22
Other Adverse Events (participants affected / at risk) | 5/23 | 5/22
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | OrthoAccel Device (N=23) | Sham (Inactive Device) (N=22)
Hypoaestesia oral (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0
Retching (Gastrointestinal disorders) | 0 | 1
Toothache (Gastrointestinal disorders) | 2 | 0
Malaise (General disorders) | 1 | 0
Sensation of pressure (General disorders) | 1 | 0
Medical device discomfort (Injury, poisoning and procedural complications) | 0 | 1
Medical device pain (Injury, poisoning and procedural complications) | 2 | 1
TAD Failure (Injury, poisoning and procedural complications) | 1 | 1
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 2
Hypoaesthesia (Nervous system disorders) | 1 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less